CLINICAL TRIAL: NCT05472935
Title: Implementing Mindfulness Based Stress Reduction Through a Learning Management System to Reduce Burnout Among Private Practice Licensed Clinical Social Workers
Brief Title: Asynchronous Mindfulness Based Stress Reduction to Reduce Burnout in Licensed Clinical Social Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Matthew L. Schwartz, Doctor of Social Work Candidate, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006599
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Burnout, Professional; Work Related Stress; Quality of Life
Keywords: Mindfulness; Mindfulness Based Stress Reduction; MBSR; Burnout; Stress Reduction; Professional Quality of Life; Social Work; Clinical Social Work; Private Practice
MeSH Terms: conditions — Burnout, Professional; Occupational Stress; Burnout, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Quasi-experimental with pre-test/post-test survey and measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBSR Intervention (Experimental): Participants will engage with MBSR instructional videos. The videos are 30 minutes in length, and designed to be watched once a day, Monday-through-Friday, over an eight-week period. Additionally, a coaching video of three minutes in length will be available to participants on Mondays. Participants will watch the videos and engage with the content and activities as prompted by the videos. Activities include guided meditations, guided mindfulness activities, such as body scans where participants notice the sensations they feel in various parts of their body, and relaxation exercises. Participants will also be asked to complete light exercises to their comfort level, which involves getting comfortable, light self-guided stretching, and relaxation exercises that are no more physical exertion than they otherwise might experience while moving around completing their normal tasks/activities of daily living outside of this program.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — Mindfulness Based Stress Reduction (MBSR) is an evidenced based intervention utilized to reduce stress.

SUMMARY:
This is a quasi-experimental study that will examine whether mindfulness based stress reduction, adapted to an online learning management system, will reduce factors related to burnout in private practice licensed clinical social workers in New York State.

DETAILED DESCRIPTION:
Mindfulness Based Stress Reduction (MBSR) is an evidenced based intervention utilized to reduce stress. In this study, MBSR is adapted as psychoeducational/instructional videos to be viewed on a learning management system by licensed clinical social workers in order to determine its efficacy in reducing symptoms related to burnout in licensed clinical social workers.

The videos are 30 minutes in length, and designed to be watched once a day, Monday-through-Friday, over an eight-week period. Additionally, a coaching video of three minutes in length will be available to participants on Mondays. Participants will watch the videos and engage with the content and activities as prompted by the videos. Activities include guided meditations, guided mindfulness activities, such as body scans where participants notice the sensations they feel in various parts of their body, and relaxation exercises. Participants will also be asked to complete light exercises to their comfort level, which involves getting comfortable, light self-guided stretching, and relaxation exercises that are no more physical exertion than they otherwise might experience while moving around completing their normal tasks/activities of daily living outside of this program.

Participants will complete a pre-test involving two validated measures, and several Likert scale, non-validated questions, and demographic questions, and a post-test, involving the same two validated measures in the pre-test (in order to determine if a statistically significant change in stress reduction has occurred) as well as completing several non-validated Likert scaling questions, and qualitative questions to determine participant's attitudes and beliefs as it relates to their participation in this research project, and their overall impression of the project elements.

ELIGIBILITY:
Inclusion Criteria:

* Licensed Clinical Social Workers in New York State
* Working in Private Practice in New York State

Exclusion Criteria:

* Anyone who does not hold a license to practice clinical social work in New York State
* Anyone who is not working in private practice as a licensed clinical social worker in New York State

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in score on the Maslach Burnout Inventory - Human Services Survey | Baseline and Week 8
  The MBI-HSS is a validated, self-reported instrument used to assess symptoms of burnout in human services workers.
Change from Baseline in score on the ProQOL 5 | Baseline and Week 8
  The ProQOL 5 (Professional Quality of Life, Version 5) Measure is a validated measure that is used for participants to self-report their overall feelings/impressions of a positive or negative professional quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Louanne Bakk, PhD, MSW, Study Chair — SUNY Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. All data will be reported in aggregate.